CLINICAL TRIAL: NCT05455047
Title: Study of Metabolic Connectivity in Drug-resistant Temporal Epilepsy
Acronym: EPINE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2021PI190
Record Dates: First submitted 2021-10-13; First posted 2022-07-13 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET-CT at 18F-FDG — PET-CT at 18f6FDG in nuclear medicine departement of Nancy's hospital

SUMMARY:
18F-Fluoro-deoxy-glucose (18F-FDG) positron emission tomography (PET) has a high sensitivity for temporal lobe epilepsy (TLE), the most common form of focal epilepsy, with a detection range of 86-90% . Therefore, 18F-FDG PET is a useful tool to identify the epileptogenic zone (ETZ) in the inter-ictal phase of drug-resistant temporal epilepsy during pre-surgical evaluation . Based on stereotactic electroencephalography (SEEG) findings, a correspondence between electrical data and metabolic changes on PET was found at the group level by identifying four different patterns of TLE . As expected, hypometabolism was not limited to the EZ defined by SEEG, but underlay broader epileptic networks . Because of the different electroclinical presentations of TLE, 18F-FDG PET appears to be a very useful tool in these temporal epilepsies. Indeed, it has been recently demonstrated that a gradient of PET hypometabolism from the uninvolved area to the spreading area, then to the epileptogenic area and to the lesion area is observed with consequently a good performance of 18F-FDG PET in defining the EZ .

Therefore, it is interesting to study PET metabolism as a network and not as a combination of regional metabolic measures in epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with drug-resistant temporal epilepsy with an accurate diagnosis on SEEG
* Patients with epilepsy who have had a PET/CT scan with 18F-FDG as part of a pre-operative assessment
* Person having received complete information on the organization of the research and not having objected to the use of these data;
* Patients affiliated to a social security system

Exclusion Criteria:

* Person who has not received full information on the organization of the research and who has opposed the use of this data
* A person of full age who is the subject of a legal protection measure (guardianship, curatorship, safeguard of justice).
* A person of full age who is unable to give consent and who is not subject to a legal protection measure

Ages: 18 Years to 56 Years | Sex: All
Age Groups: Adult
Study Population: Patients who came to the nuclear medicine department between 2009 and 2021 for an 18F-FDG PET/CT scan as part of a pre-operative assessment for epilepsy surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Metabolic connectivity | 1 month
  Metabolic connectivity of hypometabolic clusters in each temporal epilepsy subgroup defined by IRCA (interregional correlation analysis) and graph theory

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy's Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No